CLINICAL TRIAL: NCT00568841
Title: A Phase-II Clinical Trial to Evaluate the Accuracy of FDG-/FLT-PET for Early Prediction of Non-progression in Patients With Advanced NSCLC Treated With Erlotinib and to Associate PET Findings With Molecular Markers
Brief Title: Erlotinib and Sequential Positron Emission Tomography (PET) in Advanced Non Small Cell Lung Cancer (NSCLC)
Acronym: ERLOPET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lung Cancer Group Cologne (Other)
Responsible Party: Prof. Dr. Juergen Wolf, University Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2005-005393-73; 06159
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: advanced Non-Small-Cell Lung Cancer; erlotinib; FDG-PET; FLT-PET
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: erlotinib; Procedure: FDG-/FLT-PET

INTERVENTIONS:
Drug: erlotinib — erlotinib p.o. (by mouth), 150 mg once daily for week 1-6 (day 1-42)
Procedure: FDG-/FLT-PET

SUMMARY:
This is a Phase-II Study to evaluate the accuracy of Fluorodeoxyglucose-/Fluorothymidine-Positron Emission Tomography (FDG-/FLT-PET) analyses for early prediction of non-progression in patients with non-small-cell lung cancer (NSCLC) treated with Erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ≥ 18 years of age
* Untreated non-small-cell lung cancer stage IIIB/IV
* Life expectancy > 3 months
* Performance status ECOG 0-2

Exclusion Criteria:

* Concurrent systemic immune therapy, chemotherapy or therapy with any anticancer drug not indicated in the study protocol
* Any investigational agent(s) within 4 weeks prior to study entry
* Previous administration of any EGFR-targeted therapy (antibodies, small molecules and others)
* Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the accuracy of FDG-/FLT-PET analyses for early prediction of non-progression in patients with NSCLC treated with Erlotinib | 34 months

SECONDARY OUTCOMES:
To identify PET characteristics for progression, response and stable disease; To identify EGFR and KRAS sequence characteristics for clinical response and stable disease; Safety; Response rates; One-year FFTF; One-year OS; Median overall survival time | 34 months

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Wolf, Prof., Dr., Principal Investigator — University Cologne, Lung Cancer Group Cologne
Locations (1):
- Center for Integrated Oncology, University Hospital Cologne, Department I of Internal Medicine, Kerpenerstr.62, Cologne, Germany

REFERENCES:
- [Background] Barthel H, Cleij MC, Collingridge DR, Hutchinson OC, Osman S, He Q, Luthra SK, Brady F, Price PM, Aboagye EO. 3'-deoxy-3'-[18F]fluorothymidine as a new marker for monitoring tumor response to antiproliferative therapy in vivo with positron emission tomography. Cancer Res. 2003 Jul 1;63(13):3791-8. PMID 12839975
- [Background] Buck AK, Halter G, Schirrmeister H, Kotzerke J, Wurziger I, Glatting G, Mattfeldt T, Neumaier B, Reske SN, Hetzel M. Imaging proliferation in lung tumors with PET: 18F-FLT versus 18F-FDG. J Nucl Med. 2003 Sep;44(9):1426-31. PMID 12960187
- [Background] Buck AK, Schirrmeister H, Hetzel M, Von Der Heide M, Halter G, Glatting G, Mattfeldt T, Liewald F, Reske SN, Neumaier B. 3-deoxy-3-[(18)F]fluorothymidine-positron emission tomography for noninvasive assessment of proliferation in pulmonary nodules. Cancer Res. 2002 Jun 15;62(12):3331-4. PMID 12067968
- [Background] Cappuzzo F, Hirsch FR, Rossi E, Bartolini S, Ceresoli GL, Bemis L, Haney J, Witta S, Danenberg K, Domenichini I, Ludovini V, Magrini E, Gregorc V, Doglioni C, Sidoni A, Tonato M, Franklin WA, Crino L, Bunn PA Jr, Varella-Garcia M. Epidermal growth factor receptor gene and protein and gefitinib sensitivity in non-small-cell lung cancer. J Natl Cancer Inst. 2005 May 4;97(9):643-55. doi: 10.1093/jnci/dji112. PMID 15870435
- [Background] D'Addario G, Pintilie M, Leighl NB, Feld R, Cerny T, Shepherd FA. Platinum-based versus non-platinum-based chemotherapy in advanced non-small-cell lung cancer: a meta-analysis of the published literature. J Clin Oncol. 2005 May 1;23(13):2926-36. doi: 10.1200/JCO.2005.03.045. Epub 2005 Feb 22. PMID 15728229
- [Background] Fukuoka M, Yano S, Giaccone G, Tamura T, Nakagawa K, Douillard JY, Nishiwaki Y, Vansteenkiste J, Kudoh S, Rischin D, Eek R, Horai T, Noda K, Takata I, Smit E, Averbuch S, Macleod A, Feyereislova A, Dong RP, Baselga J. Multi-institutional randomized phase II trial of gefitinib for previously treated patients with advanced non-small-cell lung cancer (The IDEAL 1 Trial) [corrected]. J Clin Oncol. 2003 Jun 15;21(12):2237-46. doi: 10.1200/JCO.2003.10.038. Epub 2003 May 14. PMID 12748244
- [Background] Hanna N, Shepherd FA, Fossella FV, Pereira JR, De Marinis F, von Pawel J, Gatzemeier U, Tsao TC, Pless M, Muller T, Lim HL, Desch C, Szondy K, Gervais R, Shaharyar, Manegold C, Paul S, Paoletti P, Einhorn L, Bunn PA Jr. Randomized phase III trial of pemetrexed versus docetaxel in patients with non-small-cell lung cancer previously treated with chemotherapy. J Clin Oncol. 2004 May 1;22(9):1589-97. doi: 10.1200/JCO.2004.08.163. PMID 15117980
- [Background] Jackman DM, Yeap BY, Lindeman NI, Fidias P, Rabin MS, Temel J, Skarin AT, Meyerson M, Holmes AJ, Borras AM, Freidlin B, Ostler PA, Lucca J, Lynch TJ, Johnson BE, Janne PA. Phase II clinical trial of chemotherapy-naive patients > or = 70 years of age treated with erlotinib for advanced non-small-cell lung cancer. J Clin Oncol. 2007 Mar 1;25(7):760-6. doi: 10.1200/JCO.2006.07.5754. Epub 2007 Jan 16. PMID 17228019
- [Background] Jager PL, Gietema JA, van der Graaf WT. Imatinib mesylate for the treatment of gastrointestinal stromal tumours: best monitored with FDG PET. Nucl Med Commun. 2004 May;25(5):433-8. doi: 10.1097/00006231-200405000-00002. PMID 15100500
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Kris MG, Natale RB, Herbst RS, Lynch TJ Jr, Prager D, Belani CP, Schiller JH, Kelly K, Spiridonidis H, Sandler A, Albain KS, Cella D, Wolf MK, Averbuch SD, Ochs JJ, Kay AC. Efficacy of gefitinib, an inhibitor of the epidermal growth factor receptor tyrosine kinase, in symptomatic patients with non-small cell lung cancer: a randomized trial. JAMA. 2003 Oct 22;290(16):2149-58. doi: 10.1001/jama.290.16.2149. PMID 14570950
- [Background] Leyton J, Latigo JR, Perumal M, Dhaliwal H, He Q, Aboagye EO. Early detection of tumor response to chemotherapy by 3'-deoxy-3'-[18F]fluorothymidine positron emission tomography: the effect of cisplatin on a fibrosarcoma tumor model in vivo. Cancer Res. 2005 May 15;65(10):4202-10. doi: 10.1158/0008-5472.CAN-04-4008. PMID 15899811
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Background] Paez JG, Janne PA, Lee JC, Tracy S, Greulich H, Gabriel S, Herman P, Kaye FJ, Lindeman N, Boggon TJ, Naoki K, Sasaki H, Fujii Y, Eck MJ, Sellers WR, Johnson BE, Meyerson M. EGFR mutations in lung cancer: correlation with clinical response to gefitinib therapy. Science. 2004 Jun 4;304(5676):1497-500. doi: 10.1126/science.1099314. Epub 2004 Apr 29. PMID 15118125
- [Background] Pao W, Miller V, Zakowski M, Doherty J, Politi K, Sarkaria I, Singh B, Heelan R, Rusch V, Fulton L, Mardis E, Kupfer D, Wilson R, Kris M, Varmus H. EGF receptor gene mutations are common in lung cancers from "never smokers" and are associated with sensitivity of tumors to gefitinib and erlotinib. Proc Natl Acad Sci U S A. 2004 Sep 7;101(36):13306-11. doi: 10.1073/pnas.0405220101. Epub 2004 Aug 25. PMID 15329413
- [Background] Pao W, Miller VA, Politi KA, Riely GJ, Somwar R, Zakowski MF, Kris MG, Varmus H. Acquired resistance of lung adenocarcinomas to gefitinib or erlotinib is associated with a second mutation in the EGFR kinase domain. PLoS Med. 2005 Mar;2(3):e73. doi: 10.1371/journal.pmed.0020073. Epub 2005 Feb 22. PMID 15737014
- [Background] Perez-Soler R, Chachoua A, Hammond LA, Rowinsky EK, Huberman M, Karp D, Rigas J, Clark GM, Santabarbara P, Bonomi P. Determinants of tumor response and survival with erlotinib in patients with non--small-cell lung cancer. J Clin Oncol. 2004 Aug 15;22(16):3238-47. doi: 10.1200/JCO.2004.11.057. PMID 15310767
- [Background] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125
- [Background] Pieterman RM, van Putten JW, Meuzelaar JJ, Mooyaart EL, Vaalburg W, Koeter GH, Fidler V, Pruim J, Groen HJ. Preoperative staging of non-small-cell lung cancer with positron-emission tomography. N Engl J Med. 2000 Jul 27;343(4):254-61. doi: 10.1056/NEJM200007273430404. PMID 10911007
- [Background] Reck M, Buchholz E, Romer KS, Krutzfeldt K, Gatzemeier U, Manegold C. Gefitinib monotherapy in chemotherapy-naive patients with inoperable stage III/IV non-small-cell lung cancer. Clin Lung Cancer. 2006 May;7(6):406-11. doi: 10.3816/clc.2006.n.025. PMID 16800967
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Shepherd FA, Dancey J, Ramlau R, Mattson K, Gralla R, O'Rourke M, Levitan N, Gressot L, Vincent M, Burkes R, Coughlin S, Kim Y, Berille J. Prospective randomized trial of docetaxel versus best supportive care in patients with non-small-cell lung cancer previously treated with platinum-based chemotherapy. J Clin Oncol. 2000 May;18(10):2095-103. doi: 10.1200/JCO.2000.18.10.2095. PMID 10811675
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Spira A, Ettinger DS. Multidisciplinary management of lung cancer. N Engl J Med. 2004 Jan 22;350(4):379-92. doi: 10.1056/NEJMra035536. No abstract available. PMID 14736930
- [Background] Stroobants S, Goeminne J, Seegers M, Dimitrijevic S, Dupont P, Nuyts J, Martens M, van den Borne B, Cole P, Sciot R, Dumez H, Silberman S, Mortelmans L, van Oosterom A. 18FDG-Positron emission tomography for the early prediction of response in advanced soft tissue sarcoma treated with imatinib mesylate (Glivec). Eur J Cancer. 2003 Sep;39(14):2012-20. doi: 10.1016/s0959-8049(03)00073-x. PMID 12957455
- [Background] van Tinteren H, Hoekstra OS, Smit EF, van den Bergh JH, Schreurs AJ, Stallaert RA, van Velthoven PC, Comans EF, Diepenhorst FW, Verboom P, van Mourik JC, Postmus PE, Boers M, Teule GJ. Effectiveness of positron emission tomography in the preoperative assessment of patients with suspected non-small-cell lung cancer: the PLUS multicentre randomised trial. Lancet. 2002 Apr 20;359(9315):1388-93. doi: 10.1016/s0140-6736(02)08352-6. PMID 11978336
- [Derived] Suleiman AA, Frechen S, Scheffler M, Zander T, Kahraman D, Kobe C, Wolf J, Nogova L, Fuhr U. Modeling tumor dynamics and overall survival in advanced non-small-cell lung cancer treated with erlotinib. J Thorac Oncol. 2015 Jan;10(1):84-92. doi: 10.1097/JTO.0000000000000330. PMID 25226426
- [Derived] Scheffler M, Zander T, Nogova L, Kobe C, Kahraman D, Dietlein M, Papachristou I, Heukamp L, Buttner R, Boellaard R, Lammertsma AA, Querings S, Stoelben E, Engel-Riedel W, Neumaier B, Wolf J. Prognostic impact of [18F]fluorothymidine and [18F]fluoro-D-glucose baseline uptakes in patients with lung cancer treated first-line with erlotinib. PLoS One. 2013;8(1):e53081. doi: 10.1371/journal.pone.0053081. Epub 2013 Jan 4. PMID 23308140